CLINICAL TRIAL: NCT05821712
Title: Investigation of Clinical Efficacy of a New Mouthwash on Reducing Dental Plaque and Helping Prevent Gum Problems as Compared to a Control Mouthwash - a Six-month Study in Italy
Brief Title: A New Mouthwash on Reducing Dental Plaque and Helping Prevent Gum Problems
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CRO-2020-12-PGN-MMW-ITA-YPZ
Record Dates: First submitted 2023-03-27; First posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Plaque; Gum Disease
MeSH Terms: conditions — Plaque, Amyloid; Gingival Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 0.2% zinc lactate, 0.17% amine fluoride and 0.0275% sodium fluoride Mouthwash (Experimental): mouthwash
  Interventions: Drug: 0.2% zinc lactate, 0.17% amine fluoride and 0.0275% sodium fluoride Mouthwash
- 0.057% sodium fluoride Mouthwash (Active Comparator): mouthwash
  Interventions: Drug: 0.057% sodium fluoride Mouthwash

INTERVENTIONS:
Drug: 0.2% zinc lactate, 0.17% amine fluoride and 0.0275% sodium fluoride Mouthwash — mouthwash
  Arms: 0.2% zinc lactate, 0.17% amine fluoride and 0.0275% sodium fluoride Mouthwash
Drug: 0.057% sodium fluoride Mouthwash — mouthwash
  Arms: 0.057% sodium fluoride Mouthwash

SUMMARY:
This 6-month clinical study was designed to investigate clinical efficacy on plaque and gingivitis for the Meridol Base Mouthwash containing 0.2% zinc lactate, 0.17% amine fluoride and 0.0275% sodium fluoride as compared to a Negative Control Mouthwash containing 0.057% sodium fluoride after 3 and 6 months of product use.

ELIGIBILITY:
Inclusion Criteria:

* Subjects, ages 18-70, inclusive.
* Availability for the six-month duration of the clinical research study.
* Good general health.
* Initial gingivitis index of at least 1.0 as determined by the use of the Loe-Silness Gingival Index.
* Initial plaque index of at least 1.5 as determined by the use of the Quigley-Hein Plaque Index.
* Signed Informed Consent Form

Exclusion Criteria:

* Presence of orthodontic bands.
* Tumor(s) of the soft or hard tissues of the oral cavity.
* Advanced periodontal disease (purulent exudate, tooth mobility, and/or extensive loss of periodontal attachment or alveolar bone).
* Five or more carious lesions requiring immediate restorative treatment.
* Antibiotic use any time during the one-month period prior to entry into the study.
* Participation in any other clinical study or test panel within the one month prior to entry into the study.
* Dental prophylaxis during the past two weeks prior to baseline examinations.
* History of allergies to oral care/personal care consumer products or their ingredients.
* On any prescription medicines that might interfere with the study outcome.
* An existing medical condition that prohibits eating or drinking for periods up to 4 hours.
* History of alcohol or drug abuse.
* Self-reported pregnant or lactating subjects

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2021-09-24 (Actual); Study Completion 2021-09-24 (Actual)

PRIMARY OUTCOMES:
Gingival inflammation | baseline
  Loe-Silness Gingival Index
Gingival inflammation | 3 months
  Loe-Silness Gingival Index
Gingival inflammation | 6 months
  Loe-Silness Gingival Index

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Montesani, MD, DDS, Principal Investigator — Clinica Odontoiatrica Montesani
Locations (1):
- Clinica Odontoiatrica Montesani, Roma, Rome, Italy

REFERENCES:
- [Derived] Montesani L, Montesani L, Mateo L, Daep C, Huber N, Isapour G, Zhang YP. Antibacterial and clinical effectiveness of a mouthwash with a novel active system of amine + zinc lactate + fluoride: a randomized controlled trial. Clin Oral Investig. 2024 Jan 13;28(1):90. doi: 10.1007/s00784-023-05487-0. PMID 38217757